CLINICAL TRIAL: NCT06988072
Title: Official Title Étude Des réponses Immunes Anti-BKPyV Chez Les Patients transplantés rénaux Avec BKPyV virémie
Brief Title: Study of Anti-BKPyV Immune Responses in Kidney Transplant Patients With BKPyV Viremia
Acronym: NEPHRO-BK
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241147
Record Dates: First submitted 2025-04-04; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: BK Polyomavirus; Kidney Transplant
Keywords: Polyomavirus hominis 1; Natural killer cells; T-lymphocytes; Neutralizing antibodies; Adaptative immunity; Immunologic memory; Innate immunity recognition; Trained immunity; Immune repertoire; Biomarkers; BKPyV-association nephropathy
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Kidney transplant recipients with de novo BKPyV DNAemia: kidney transplant recipients with de novo BKPyV DNAemia within the first 12 months post-transplantation, including adult and pediatric patients
  Interventions: Other: blood sampling
- Control subjects : Healthy adult donors from the National blood bak
  Interventions: Other: blood sampling
- Control subjects : Kidney transplant recipients without BKPyV DNAemia
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — At BKPyV reactivation, at 1 month, 3 months and 12 months
  Groups: Kidney transplant recipients with de novo BKPyV DNAemia
Other: blood sampling — once
  Groups: Control subjects : Healthy adult donors from the National blood bak
Other: blood sampling — once
  Groups: Control subjects : Kidney transplant recipients without BKPyV DNAemia

SUMMARY:
The human pathogen BK polyomavirus (BKPyV) is a ubiquitous, small, non-enveloped DNA virus that infects over 90% of people, typically in childhood with mild or no symptoms. Following primary infection, BKPyV establishes latency predominantly in the reno-urinary tract, and can occasionally be detected in the urine without any concomitant clinical symptoms. However, among kidney transplant recipients (KTR), due to impaired cellular and humoral immunity, uncontrolled viral replication in renal tubular epithelial cells (RPTE) can occur, leading to high-level BKPyV DNAemia and significant damage to the reno-urinary system (ie polyomavirus-associated nephropathy). In the absence of any effective antiviral drug, the mainstay of therapy for significant BKPyV replication among KTR is reducing immunosuppressive drugs, despite the subsequent of risk of graft rejection. Current efforts to identify new monitoring and therapeutical strategies need to be supported by a better understanding of the dynamics of BKPyV-specific immune responses following transplantation.

Although adaptive cellular and humoral immune responses play a crucial role in the control of BKPyV reactivation among healthy individuals, immunosuppression and transplantation disrupt immune homeostasis and reshape the immune response landscape both in terms of function and fitness to new stimuli. Consequently, pre-transplant prediction of patients who will be able to control post-transplant BKPyV reactivation or who will develop BKPyV-related complications remains challenging. This knowledge gap stems from insufficient studies on the comprehensive analysis of immune responses during BKPyV reactivation. In particular, most studies to date have not investigated the role of NK cells in this context, despite their potent antiviral activity, heterogenous repertoire in each patient and their recently uncovered adaptive properties.

The hypothesis is that among KTR with de novo BKPyV DNAemia, the comprehensive analysis of anti-BKPyV immune responses (including both the description of NK cell repertoire and adaptive immune), could allow

* A better stratification of KTR at-risk for BKPyV-related complications using accessible immune biomarkers.
* The identification of the most efficient strategies of immunosuppression management for the control of BKPyV DNAemia, that could be further evaluated in a prospective cohort.
* The identification of immunological correlates for the control of BKPyV DNAemia, which aim at providing a foundation for the development of future immunotherapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* No objection to participation in the research study (from patients or legal guardians)
* Affiliated to the French national social security system
* Age ≥ 7 years old
* Weight ≥ 12 kg

Additional criteria for kidney transplant recipients with BKPyV DNAemia:

* Patients who underwent kidney transplantation within 12 months prior to inclusion, regardless of the initial indication
* Detectable de novo BKPyV DNAemia within the first 12 months post-transplantation

Additional criteria for kidney transplant recipients without BKPyV DNAemia:

* Patients who underwent kidney transplantation within 12 months prior to inclusion, regardless of the initial indication
* No detectable de novo BKPyV DNAemia within the first 12 months post-transplantation

Additional criteria for healthy donors (controls):

* Age ≥ 18 years old
* Blood donation to the EFS
* Consent for the use of their blood donation for research purposes.

Exclusion Criteria:

* Objection to participation in the research study

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population: kidney transplant recipients with de novo BKPyV DNAemia within the first 12 months post-transplantation, including adult and pediatric patients.
  Control subjects: control subjects will be matched to the study patients (criteria below with a ratio of 1-1-1):
  * Healthy adult donors from the National blood bak (Etablissement Français du Sang - EFS): these control patients will be matched to study population patients on age (± 5ans) and sex
  * Kidney transplant recipients without BKPyV DNAemia, enrolled within the active cohorts of the participating centers: these control patients will be matched to study population patients on age (± 5ans), enrolling center, time since transplantation (± 3 months), and sex.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of circulating NK cells | At inclusion
  NK cells circulating repertoire defects associated with BKPyV-DNAemia Extensive characterization of the phenotype of circulating NK cells among kidney transplant recipients with de novo BKPyV DNAemia to predict the clinically relevant outcome "BKPyV reactivation control"
Number of circulating NK cells | At 1 month
  NK cells circulating repertoire defects associated with BKPyV-DNAemia Extensive characterization of the phenotype of circulating NK cells among kidney transplant recipients with de novo BKPyV DNAemia to predict the clinically relevant outcome "BKPyV reactivation control"
Number of circulating NK cells | At 3 months
  NK cells circulating repertoire defects associated with BKPyV-DNAemia Extensive characterization of the phenotype of circulating NK cells among kidney transplant recipients with de novo BKPyV DNAemia to predict the clinically relevant outcome "BKPyV reactivation control"
Number of circulating NK cells | At 12 months
  NK cells circulating repertoire defects associated with BKPyV-DNAemia Extensive characterization of the phenotype of circulating NK cells among kidney transplant recipients with de novo BKPyV DNAemia to predict the clinically relevant outcome "BKPyV reactivation control"

SECONDARY OUTCOMES:
Frequency of Functional Impact of BKPyV Reactivation on NK Cell Effector Functions | Up to 12 months
  Cytotoxicity assays of NK cells in response to antigenic stimulation (pre-specified BKPyV peptides) and co-culture models (BKPyV-infected RPTEC) At each available timepoint
Frequency of T- and B-cell specific functional responses in patients with de novo BKPyV reactivation | Up to 12 months
  Viral neutralization assays (humoral responses) and anti-BKPyV ELISPOT assays (T cell responses) At each available timepoint
Correlation between the main changes in immunosuppressive treatment and the anti-BPyV immune response | Up to 12 months
  Correlation between the main changes in immunosuppressive treatment carried out after the appearance and BKPyV viremia and the anti-BKPyV immune response assessed by the immunological biomarkers
Correlation between the main changes in immunosuppressive treatment and the control of BKPyV viremia | Up to 12 months
Correlation between the main changes in immunosuppressive treatment and the occurrence of BKPyV nephropathy | Up to 12 months
Correlation between the main changes in immunosuppressive treatment and the occurrence of rejection | Up to 12 months
BKPyV viral diversity evolution during clinical course of infection | Up to 12 months
  Whole genome sequencing (WGS) of BKPyV on consecutive plasma sample among patients with BKPyV DNAemia (characterization of major and minor viral subpopulations, identification of coinfections) At eaxh available timetpoint
Impact of BKPyV reactivation on alloreactive properties of NK cells | Up to 12 months
  NK cells cytotoxicity assessments against allogenic endothelial cells after stimulation by BKPyV (infected cells and/or BKPyV isolated peptides)

IPD SHARING:
Plan to Share IPD: Undecided